CLINICAL TRIAL: NCT03762382
Title: Phase IIa, 90-Day Safety, Adherence, and Acceptability Study of Intravaginal Rings Releasing Tenofovir With and Without Levonorgestrel Among Women in Western Kenya
Brief Title: Tenofovir/Levonorgestrel Intravaginal Ring and Tenofovir Intravaginal Ring
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: CONRAD (Other)
Collaborators: Kenya Medical Research Institute (Other); University of Washington (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Protocol B17-144; RFA-PS-17-005 (Other Grant/Funding Number: U.S. Centers for Disease Control and Prevention); AID-OAA-A-14-000010 (Other Grant/Funding Number: USAID)
Record Dates: First submitted 2018-11-16; First posted 2018-12-03 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: HIV; Contraception; Prevention; Anti-Retroviral Agent
Keywords: Intravaginal Ring; HIV Prevention; Tenofovir; Levonorgestrel; Pregnancy Prevention
MeSH Terms: interventions — Tenofovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TFV/LNG IVR (10mg/20μg) (Continuous) (Experimental): Tenofovir/Levonorgestrel Intravaginal Ring
  Interventions: Drug: TFV/LNG IVR
- TFV IVR (10mg) (Continuous) (Experimental): Tenofovir Intravaginal Ring
  Interventions: Drug: TFV IVR
- Placebo IVR (Non-eluting) (Placebo Comparator): Placebo Intravaginal Ring
  Interventions: Drug: Placebo IVR

INTERVENTIONS:
Drug: TFV/LNG IVR — TFV/LNG IVR is an intravaginal ring that releases approximately 8-10 mg/day of TFV and approximately 20ug/day of LNG to be used for 90 continuous days.
  Other Names: Tenofovir/Levonorgestrel Intravaginal Ring
  Arms: TFV/LNG IVR (10mg/20μg) (Continuous)
Drug: TFV IVR — TFV IVR is an intravaginal ring that releases approximately 8-10mg/day of TFV to be used for 90 continuous days.
  Other Names: Tenofovir Intravaginal Ring
  Arms: TFV IVR (10mg) (Continuous)
Drug: Placebo IVR — Placebo IVR is an intravaginal ring containing no active experimental ingredients to be used for 90 continuous days.
  Arms: Placebo IVR (Non-eluting)

SUMMARY:
The purpose of the study is to evaluate the safety, pharmacokinetics and pharmacodynamics of, and the tolerability and acceptance of an intravaginal ring (IVR) delivering both tenofovir and levonorgestrel (TFV/LNG) and an IVR delivering TFV only, compared to a placebo IVR, in women in Western Kenya.

DETAILED DESCRIPTION:
This Phase 2a clinical trial will evaluate the safety, pharmacokinetics and pharmacodynamics of, and the tolerability and adherence to two novel intravaginal rings (IVRs). The tenofovir/levonorgestrel (TFV/LNG) IVR and TFV IVRs are designed to provide HIV (and HSV-2) prevention with and without contraceptive for pregnancy prevention, respectively. Women will be protected from pregnancy by abstinence from vaginal intercourse or agreeing to consistently use condoms; concurrent use of a non-hormonal copper intrauterine device is permitted.

The study will enroll healthy, HIV-negative, non-pregnant, menstruating women aged 18-34 years, inclusive, and not currently infected with hepatitis B virus, who are assessed to be at lower risk for HIV. The goal is to enroll fifty (50) women in Western Kenya. The participants will be randomized 2:2:1 to use one of the following continuous delivery IVRs: twenty (20) women to use the TFV/LNG IVR; ten (10) women to use the TFV IVR; and ten (10) women to use the placebo IVR. Participants will attend up to ten (10) routine study visits that may include physical and pelvic exams, collection of venous blood, vaginal fluid and cervical mucus, and behavioral questionnaires. A subset of twenty (20) women will participate in in-depth interviews.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged 18-34 years, inclusive
* General good health (by history and per clinician discretion) without any clinically significant systemic disease (including, but not limited to significant liver disease/hepatitis, gastrointestinal disease, kidney disease, thyroid disease, osteoporosis or bone disease, and diabetes), uterus, and cervix
* Not pregnant or planning to become pregnant
* Pre-screening HIV risk score ≤4
* Currently having regular menstrual cycles (approximately 24-35 days) OR with a history of having regular menstrual cycles before contraceptive use, by report, and resumed some menstruation or spotting (with biochemical confirmation of ovulation)
* Willing to undergo Visual Inspection with Lugol's Iodine (VILI) for cervical abnormalities during pelvic exam
* Willing to abstain from use of vaginal products other than the study product, including tampons (except for during menses) , menstrual cups, vaginally inserted cloths or other materials, spermicides, lubricants, and douches for the whole study
* Willing to abstain from any vaginal intercourse starting 48 hours before certain study visits
* Vaginal and cervical anatomy that, in the opinion of the clinician, lends itself to easy genital tract sample collection and is absent of vesicles and ulcers
* No use of hormonal contraceptives within the following periods specified for each type of contraception method:

  * Oral contraceptives (combined or progestin-only), contraceptive patch or contraceptive vaginal ring in at least two (2) months
  * Last DMPA injection received at least four (4) months ago and has resumed regular menstruation
  * Hormonal IUD/IUS removed at least four (4) months ago and has resumed regular menstruation
  * Hormonal implant removed at least six (6) months ago and has resumed regular menstruation
* Willing to refrain from using any hormonal contraceptives for the entire study and to use only study-provided non-spermicidal male condoms with or without a study-provided Cu-IUD
* P4 ≥3.0 ng/ml
* Estimated glomerular filtration rate (eGFR) ≥90ml/min/1.73m2
* Willing to give voluntary consent and sign/mark an informed consent form
* Willing and able to comply with protocol requirements

Exclusion Criteria:

* Body mass index (BMI) ≥30 kg/m
* History of hysterectomy
* Currently pregnant or within less than three (3) calendar months of the last pregnancy outcome.
* Currently breastfeeding or having breastfed an infant in the last two (2) months, or planning to breastfeed during the course of the study
* Contraindication to any study products-LNG, TFV, or excipient ingredients
* Contraindication to LNG
* In the last three (3) months, diagnosed with or treated for any STI or pelvic inflammatory disease
* Positive test for HIV-1, syphilis, Trichomonas vaginalis (TV), Neisseria gonorrhea (GC), Chlamydia trachomatis (CT) or HBsAg
* Nugent score greater than or equal to 7 or a symptomatic BV clinical diagnosis as defined by Amsel's criteria
* Suspected breast cancer or other progestin-sensitive cancer
* Suspected hepatic disease, including cirrhosis or viral hepatitis
* History of bleeding or coagulation problems
* Known current drug or alcohol abuse which could impact study compliance
* Grade 2 or higher laboratory abnormality, per the Division of AIDS, National Institute of Allergy and Infectious Disease (DAIDS) Table for Grading the Severity of Adverse Events, or clinically significant laboratory abnormality as determined by the clinician
* Use of any concomitant medications
* Participation in any other investigational trial with use of a drug/device within the last 30 days or planned participation in any other investigational trial with use of a drug/device during the study
* History of gynecological procedures (including genital piercing) on the external genitalia, vagina, or cervix within the last 14 days
* Labial elongation (due to pulling practices and use of botanicals or caustic agents)
* Abnormal finding on laboratory or physical examination or a social or medical condition in the volunteer which, in the opinion of the site co-PI(s), would make participation in the study unsafe or would complicate interpretation of data
* Currently using, or has used within the preceding one (1) month, emtricitabine/tenofovir disoproxil fumarate (TDF/FTC or Truvada®) or any other tenofovir product, and/or has plans to use a non-study tenofovir product in any form during the study

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy, non-pregnant females of reproductive potential, ovulating and not using non-study hormonal contraception during the study period.
Enrollment: 50 (Estimated)
Dates: Start 2018-12-12 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Treatment-emergent adverse events (TEAEs) | Change from Baseline to up to 90 days of IVR use
  Participants with Grade 2 or higher local female genital TEAEs as defined by DAIDS Table for Grading the Severity of Adult and Pediatric AEs (version 2.1) and DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events Addendum 1 Female Genital Grading Table for Use in Microbicide Studies
Safety Laboratory Assessments- Serum chemistry | Change from Baseline to up to 90 days of IVR use
  Number of participants with abnormal serum chemistry
Safety Laboratory Assessments- lipids | Change from Baseline to up to 90 days of IVR use
  Number of participants with abnormal lipids
Safety Laboratory Assessments- complete blood counts | Change from Baseline to up to 90 days of IVR use
  Number of participants with abnormal complete blood counts
Mucosal safety | Change from Baseline to up to 90 days of IVR use
  Changes in cervicovaginal mucosa by visual inspection

SECONDARY OUTCOMES:
Maximum blood concentrations (Cmax) | Baseline; 6 and 24 hours post IVR insertion; Menstrual cycle 1, day 14; Menstrual cycle 1,day 21-25; Menstrual cycle 2, day 21-25; Menstrual cycle 3, day 14; Day 90 IVR use; 24 hours post-IVR use (anticipated cycle length is 28 days)
  Maximum plasma concentration of TFV and maximum serum concentration of LNG
Maximum CV fluid concentration | 6 and 24 hours post-IVR insertion; Menstrual cycle 1 day 14; Menstrual cycle 1 day 21-25; Menstrual cycle 2 day 21-25; Menstrual cycle 3, day 14; Day 90 of IVR use; and 24 hours post-IVR use (anticipated cycle length is 28 days)
  Maximum CV fluid concentration of TFV
Percent (%) inhibition of HIV resulting from product use (Anti-HIV activity) | Baseline, Day 90 of IVR use
  Anti-HIV and anti-HSV-2 activity in CV fluid (inhibition in cell assay)
Percent (%) inhibition of HSV resulting from product use (Anti-HSV activity) | Baseline, Day 90 of IVR use
  Anti-HSV-2 activity in CV fluid (inhibition in cell assay)
Cervical mucus assessment and quality score | Menstrual cycle 1, day 14; Menstrual cycle 3, day 14 (anticipated cycle length is 28 days)
  Cervical mucus assessment and quality score (total summary score 0-15) as defined by WHO laboratory manual for the Examination and processing of human semen Fifth Edition, Appendix 5
Confirmation of Ovulation | Pre-IVR insertion; Menstrual cycle 1, day 20-25; Menstrual cycle 2, day 20-25; Day 90 of IVR use (anticipated cycle length is 28 days)
  Serum progesterone (P4) level.
Cervicovaginal (CV) fluid cytokines-IL-1α | Change from Baseline to Day 90 of IVR use
  Changes in IL-1α in CV fluid.
Cervicovaginal (CV) fluid cytokines- IL-8 | Change from Baseline to Day 90 of IVR use
  Changes in IL-8 in CV fluid.
Changes in endogenous vaginal bacteria | Change from Baseline to Day 90 of IVR use
  Changes in endogenous vaginal bacteria in CV fluid
Changes in endogenous vaginal bacteria- Nugent score | Change from Baseline to Day 90 of IVR use
  Changes in Nugent score (score 0-10)
qPCR of Ring Microbiota | Day 90 of IVR use
  Microbial growth on returned IVRs.
Tolerability - Somatic and non-specific non-treatment emergent adverse events | Baseline; 6 and 24 hours post-IVR insertion; Menstrual cycle 1, day 14; Menstrual cycle 1, day 21-25; Menstrual cycle 2, day 21-25; Menstrual cycle 3, day 14; 90 days of IVR use; 24 hours post IVR use (anticipated cycle length is 28 days)
  Subjective and objective assessment of new complaints (e.g., headache, nausea, weight change, breast tenderness, etc.)
Tolerability - Self-reported complaints of changes in menstrual cycle | Screening; Menstrual cycle 1, day 14; Menstrual cycle 1, day 21-25; Menstrual cycle 2, day 21-25; Menstrual cycle 3, day 14; Day 90 of IVR use; 24 hours post-IVR use (anticipated cycle length is 28 days)
  Percentage of women with changes in regularity of menstrual cycle
Adherence - Drug concentrations | Baseline; 6 and 24 hours post-IVR insertion; Menstrual cycle 1, day 14; Menstrual cycle 1, day 21-25; Menstrual cycle 2, day 21-25; Menstrual cycle 3, day 14; 90 days of IVR use; 24 hours post-IVR use (anticipated cycle length is 28 days)
  Plasma, serum, and vaginal fluid drug concentrations.
Adherence - Residual drug concentrations | Day 90 of IVR use
  Residual drug (TFV and LNG) concentrations in returned TFV/LNG and TFV IVRs and residual excipients in returned placebo IVRs.
Adherence - Percentage of discontinuations | Up to Day 90 of IVR use
  Percentage of IVR discontinuations
Acceptability - Quantitative assessment of acceptability based on Questionnaires administered pre- and post-IVR use | Screening; 90 days of IVR use
  Changes in responses to questionnaires pre- and post-IVR use on attitudes toward and perspectives of IVR use.

OTHER OUTCOMES:
Qualitative assessment of acceptability and adherence influences through In-depth interviews | Between Menstrual cycle 2, day 21-25 and Menstrual cycle 3, day 14 (anticipated cycle length is 28 days)
  In-depth interviews

CONTACTS AND LOCATIONS:
Overall Officials: Nelly R. Mugo, MBChB, Principal Investigator — University of Washington
Locations (1):
- Kenya Medical Research Institute, Center for Global Health Research, Kisumu, Kisumu County, Kenya

IPD SHARING:
Plan to Share IPD: No
Data sharing will comply with CDC's current Policy on Public Health Research and Non-research Data Management and Access. Except for the analyses outlined in the study protocol, all future requests to perform new analyses on data or specimens from this study protocol will require (1) agreement of all Parties owning or jointly owning the data and (2) Ethics Committee approval.

REFERENCES:
- [Background] Thurman AR, Schwartz JL, Brache V, Clark MR, McCormick T, Chandra N, Marzinke MA, Stanczyk FZ, Dezzutti CS, Hillier SL, Herold BC, Fichorova R, Asin SN, Rollenhagen C, Weiner D, Kiser P, Doncel GF. Randomized, placebo controlled phase I trial of safety, pharmacokinetics, pharmacodynamics and acceptability of tenofovir and tenofovir plus levonorgestrel vaginal rings in women. PLoS One. 2018 Jun 28;13(6):e0199778. doi: 10.1371/journal.pone.0199778. eCollection 2018. PMID 29953547
- [Derived] Mugo NR, Mudhune V, Heffron R, Thomas KK, McLellan-Lemal E, Njoroge B, Peacock S, O'Connor SM, Nyagol B, Ouma E, Ridzon R, Wiener J, Isoherranen N, Erikson DW, Ouattara LA, Yousefieh N, Jacot TA, Haaland RE, Morrison SA, Haugen HS, Thurman AR, Allen SA, Baeten JM, Samandari T, Doncel GF. Randomized controlled phase IIa clinical trial of safety, pharmacokinetics and pharmacodynamics of tenofovir and tenofovir plus levonorgestrel releasing intravaginal rings used by women in Kenya. Front Reprod Health. 2023 Jun 13;5:1118030. doi: 10.3389/frph.2023.1118030. eCollection 2023. PMID 37383290
- [Derived] McLellan-Lemal E, Deaton SR, Betts JE, Ondenge K, Mudhune V, O'Connor SM, Nyagol B, Thurman AR, Doncel GF, Allen SA, Heffron R, Mugo NR; Kisumu Combined Ring Study (KCRS) Team. Acceptability of an intravaginal ring for simultaneously preventing HIV infection and pregnancy: Qualitative findings of the Kisumu Combined Ring Study, 2019. Contemp Clin Trials. 2022 Nov;122:106935. doi: 10.1016/j.cct.2022.106935. Epub 2022 Sep 23. PMID 36162740
- [Derived] Dabee S, Mugo N, Mudhune V, McLellan-Lemal E, Peacock S, O'Connor S, Njoroge B, Nyagol B, Thurman AR, Ouma E, Ridzon R, Wiener J, Haugen HS, Gasper M, Feng C, Allen SA, Doncel GF, Jaspan HB, Heffron R; Kisumu Combined Ring Study Team. Genital microbiota of women using a 90 day tenofovir or tenofovir and levonorgestrel intravaginal ring in a placebo controlled randomized safety trial in Kenya. Sci Rep. 2022 Jul 14;12(1):12040. doi: 10.1038/s41598-022-13475-9. PMID 35835755